CLINICAL TRIAL: NCT02925793
Title: A Randomised, Double-blind, Vehicle-Controlled, Phase IIb Study to Assess the Efficacy and Safety of Topically Applied DS107 Cream to Adults With Mild to Moderate Atopic Dermatitis
Brief Title: Safety and Efficacy Study of Topically Applied DS107 Cream in Mild to Moderate Atopic Dermatitis Patients (AD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DS Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DS107E-06
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Results first posted 2022-10-07 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vehicle Cream (Placebo Comparator): Vehicle cream applied topically to all affected or commonly affected areas twice-daily for 8 weeks
  Interventions: Other: Vehicle cream
- 1% DS107 Cream (Experimental): 1% DS107 cream applied topically to all affected or commonly affected areas twice-daily for 8 weeks
  Interventions: Drug: DS107
- 5% DS107 Cream (Experimental): 5% DS107 cream applied topically to all affected or commonly affected areas twice-daily for 8 weeks
  Interventions: Drug: DS107

INTERVENTIONS:
Drug: DS107
  Other Names: 1%w/w DS107 DGLA Cream & 5%w/w DS107 DGLA Cream
  Arms: 1% DS107 Cream; 5% DS107 Cream
Other: Vehicle cream
  Other Names: DS107 Placebo Cream
  Arms: Vehicle Cream

SUMMARY:
The purpose of this randomized, double blind, placebo controlled, parallel group study is to compare the safety and efficacy of topically applied DS107 cream (1% and 5%) versus vehicle cream, in the treatment of adult patients with mild to moderate Atopic Dermatitis (AD).

DETAILED DESCRIPTION:
This was a randomized, vehicle-controlled, double-blind, parallel-group, multicenter, Phase 2b study to investigate the safety and efficacy of topically administered DS107 cream and the dose-response relationship between DS107 cream and vehicle cream in patients 18 years and older with mild to moderate AD.

Approximately 300 patients (100 per treatment group), with mild to moderate AD were to be included in this study. All patients signed the patient information sheet (PIS)/informed consent form (ICF) and underwent screening for study eligibility. Eligible patients were randomized (1:1:1) to receive 1% DS107 cream, 5% DS107 cream or, vehicle cream:

Treatment Group A: 1% DS107 cream Treatment Group B: 5% DS107 cream Treatment Group C: Vehicle cream Study cream was to be applied topically to all affected or commonly affected areas twice daily (BID) for 8 weeks. To maintain the double-blind conditions, the DS107 and vehicle creams were identical in appearance. During their participation, patients were to come to the clinic on 7 occasions: Screening, Baseline, and at Weeks 2, 4, 6, 8 (end of treatment), and 10 (follow-up).

At the start of the study, areas for treatment were defined, DS107 or vehicle cream was then applied to those areas (and any newly affected areas) throughout the 8-week treatment period. Patients were instructed to apply the study cream liberally to the affected area in the morning and the evening. Emollients could be applied to other areas of dry skin that were not in the defined treatment area. On the days of clinic visits, patients were instructed to abstain from applying study cream for 6 hours prior to the visit and then to apply study cream as soon as possible after the clinic visit.

Once enrolled, patients were restricted from using any other treatment for AD. Any medication (prescription and over-the-counter [OTC] drugs) or therapeutic intervention deemed necessary for the patient, and which in the opinion of the investigator did not interfere with the safety and efficacy evaluations, could be continued unless they were included in the prohibited list of medications and therapeutic regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinically confirmed diagnosis of active Atopic Dermatitis according to Hanifin and Rajka criteria
* Patients with mild to moderate Atopic Dermatitis at baseline as defined by an Investigator's Global Assessment (IGA) score of 3 or 2 at baseline visit
* Patients with Atopic Dermatitis covering a minimum 5% of the body surface area at baseline
* Male or female patients aged 18 years and older on the day of signing the informed consent form (ICF)

Exclusion Criteria:

* Patients with other skin conditions that might interfere with Atopic Dermatitis diagnosis and/or evaluation (such as psoriasis or current active viral, bacterial and fungal topical skin infections) as assessed by the Investigator
* Patients who have used systemic treatments (other than biologics) that could affect Atopic Dermatitis less that 4 weeks prior to baseline visit (Day 0), e.g. retinoids, methotrexate, cyclosporine, hydroxycarbamide (hydroxyurea), azathioprine and oral/injectable corticosteroids. Intranasal corticosteroids for stable medical conditions are allowed
* Patients who have used any topical medicated treatment for Atopic Dermatitis two weeks prior to the start of treatment/baseline (Day 0) including but not limited to, topical corticosteroids, calcineurin inhibitors, tars, bleach, antimicrobials, and bleach baths
* Patients who use topical products containing urea, ceramides or hyaluronic acid two weeks prior to Day 0
* Patients who have a history of hypersensitivity to any substance in DS107 cream or vehicle cream
* Patients who have any clinically significant controlled or uncontrolled medical condition or laboratory abnormality that would, in the opinion of the Investigator, put the patient at undue risk or interfere with the interpretation of study results
* Patients with significant uncontrolled cardiovascular, neurologic, malignant, psychiatric, respiratory or hypertensive disease, as well as uncontrolled diabetes and floride arthritis or any other illness that, in the opinion of the Investigator, is likely to interfere with completion of the study
* Patients with chronic infectious diseases (e.g. hepatitis B, hepatitis C, or infection with human immunodeficiency virus)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Weissbach, MD, Ph.D, Study Chair — DS Biopharma
Locations (3):
- DS Biopharma Site, East Windsor, New Jersey, United States
- DS Biopharma Site, Markham, Canada
- DS Biopharma Site, Cape Town, South Africa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 300 patients (100 per treatment group), with mild to moderate Atopic Dermatitis (AD) were to be included in this study.
Pre-assignment Details: Eligible patients were randomized (1:1:1) to receive either 1% DS107 cream, 5% DS107 cream or, vehicle cream.
Groups:
- Vehicle Cream: Vehicle cream applied topically to all affected or commonly affected areas twice-daily for 8 weeks
  Vehicle cream
- 1% DS107 Cream: 1% DS107 cream applied topically to all affected or commonly affected areas twice-daily for 8 weeks
  DS107
- 5% DS107 Cream: 5% DS107 cream applied topically to all affected or commonly affected areas twice-daily for 8 weeks
  DS107
Period: Overall Study
Arm/Group | Vehicle Cream | 1% DS107 Cream | 5% DS107 Cream
Started | 106 | 110 | 111
Completed | 81 | 81 | 83
Not Completed | 25 | 29 | 28
Not completed — Adverse Event | 3 | 3 | 6
Not completed — Withdrawal by Subject | 16 | 15 | 13
Not completed — Investigator Discretion | 0 | 1 | 1
Not completed — Lost to Follow-up | 2 | 3 | 1
Not completed — Lack of Efficacy | 2 | 6 | 4
Not completed — Other: | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All patients who were randomized to the study and received at least one dose of study cream. FAS was the primary analysis population for efficacy endpoints.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle Cream | 1% DS107 Cream | 5% DS107 Cream | Total
Number analyzed (Participants) | 106 | 110 | 110 | 326
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (16.54) | 38.2 (15.13) | 43.2 (16.06) | 40.6 (15.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 75 | 50 | 188
  Male | 43 | 35 | 60 | 138
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 16 | 23 | 22 | 61
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 1 | 5
  Black or African American | 19 | 25 | 28 | 72
  White | 55 | 48 | 50 | 153
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 15 | 11 | 9 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Numeric Rating Scale (NRS) for Pruritus in Treated Population Compared to Vehicle Population at Week 8
Description: Change from baseline in Numeric Rating Scale (NRS) for Pruritus in treated population compared to vehicle population at Week 8. Severity of pruritus related to atopic dermatitis (AD) was self-assessed by patients daily using the NRS. Patients were asked to estimate the intensity of pruritus at its worst over the previous 24 hours. The Pruritus NRS is a single-question assessment tool that was used to assess the patient's worst itch as a result of AD in the previous 24 hours. Patients scored their pruritus due to AD on a scale of 0 - 10, with 0 indicating no itch and 10 indicating the worst itch imaginable. Patients were required to complete the rating scale daily starting at screening through to the last study visit. A decrease in worst itch NRS indicates a positive outcome for the participant.
Time Frame: Baseline and Week 8
Population: The Full Analysis Set (FAS) includes all randomised patients who received at least one administration of study treatment and have at least one post-baseline measurement.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle Cream | 1% DS107 Cream | 5% DS107 Cream
Number analyzed (Participants) | 72 | 74 | 77
score on a scale | -3.8 (2.66) | -2.9 (2.66) | -2.9 (2.31)
Statistical Analysis 1: Comparison: Vehicle Cream vs 1% DS107 Cream; Both 1% and 5% groups (statistical analysis 2) produced the same estimated value (-2.9); Test type: Superiority; p = 0.0106, SAS Proc Mixed; Mean Difference = -2.9 — For each subject, change in NRS score from baseline to week 8 was calculated as Week 8 NRS value minus Baseline NRS value. Mean change in NRS score from baseline to week 8 for each group was then calculated using a Generalized Linear Mixed Model
Statistical Analysis 2: Comparison: Vehicle Cream vs 5% DS107 Cream; Both 1%(statistical analysis 1) and 5% groups produced the same estimated value (-2.9); Test type: Superiority; p = 0.0483, SAS Proc Mixed; Mean Difference = -2.9 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Change From Baseline in Eczema Area and Severity Index (EASI) in Treated Population Compared to Vehicle Population at Week 8
Description: Change from baseline in EASI in treated population compared to vehicle population at Week 8. EASI quantifies the severity of a patient's atopic dermatitis (AD) based on both lesion severity and the percent of body surface area (BSA) affected. The EASI is a composite score ranging from 0-72 that takes into account the degree of erythema, induration/papulation, excoriation, and lichenification (each scored from 0 to 3 separately, half points are permitted) for each of four body regions, with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The severity of each sign is assessed using a 4-point scale (half points are permitted):
  * 0 = none
  * 1 = mild
  * 2 = moderate
  * 3 = severe A decrease in EASI indicates a positive outcome for the participant.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle Cream | 1% DS107 Cream | 5% DS107 Cream
Number analyzed (Participants) | 80 | 80 | 83
score on a scale | -7.96 (8.504) | -7.26 (7.287) | -8.44 (7.603)

3. Secondary Outcome: Change From Baseline in NRS for Pruritus Intreated Populations Compared to Vehicle Population at Week 2, 4, 6, 10
Description: Change from baseline in NRS for Pruritus in the treated populations compared to vehicle population at Weeks 2, 4, 6, 10. Severity of pruritus related to atopic dermatitis (AD) was self-assessed by patients daily using the NRS. Patients were asked to estimate the intensity of pruritus at its worst over the previous 24 hours. The Pruritus NRS is a single-question assessment tool that was used to assess the patient's worst itch as a result of AD in the previous 24 hours. Patients will score their pruritus due to AD on a scale of 0 - 10, with 0 indicating no itch and 10 indicating the worst itch imaginable. Patients were asked to complete the rating scale daily starting at screening through to the last study visit. A decrease in worst itch NRS indicates a positive outcome for the participant.
Time Frame: Baseline, Week 2, Week 6 and Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle Cream | 1% DS107 Cream | 5% DS107 Cream
Number analyzed (Participants) | 106 | 110 | 110
score on a scale
  Week 2 | -1.5 (1.88) | -1.1 (1.68) | -1.4 (1.92)
  Week 4 | -2.7 (1.99) | -2.1 (2.45) | -2.1 (1.95)
  Week 8 | -3.3 (2.44) | -2.7 (2.61) | -2.5 (2.08)
  Week 10 | -3.8 (2.74) | -2.9 (2.90) | -3.0 (2.46)

4. Secondary Outcome: Proportion of Patients Achieving a Decrease of at Least 2.7 Points in NRS in the Treated Populations Compared to Vehicle Population From Baseline to Weeks 2, 4, 6, 8, and 10.
Description: • Proportion of Patients Achieving a Decrease of at Least 2.7 Points in Numeric Rating Scale (NRS) in Treated Population Compared to Vehicle Population from Baseline to Week 2, 4, 6, 8 and 10. The NRS for Pruritus is a single-question assessment tool that was used to assess the patient's worst itch as a result of AD in the previous 24 hours. Patients were asked to estimate the intensity of pruritus at its worst over the previous 24 hours. Patients were to score their pruritus due to AD on a scale of 0-10, with 0 (no itch) and 10 (worst itch imaginable)
Time Frame: 10 weeks
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Vehicle Cream | 1% DS107 Cream | 5% DS107 Cream
Number analyzed (Participants) | 106 | 110 | 110
Proportion of participants
  Week 2 | 0.19 | 0.14 | 0.15
  Week 4 | 0.38 | 0.26 | 0.28
  Week 6 | 0.41 | 0.31 | 0.39
  Week 8 | 0.45 | 0.31 | 0.4
  Week 10 | 0.42 | 0.31 | 0.35

5. Secondary Outcome: Change From Baseline in EASI in Treated Population Compared to Vehicle Population at Weeks 2, 4, 6, 10.
Description: Change from baseline in EASI in the treated populations compared to vehicle population at Weeks 2, 4, 6, 10. EASI quantifies the severity of a patient's atopic dermatitis (AD) based on both lesion severity and the percent of body surface area (BSA) affected. The EASI is a composite score ranging from 0-72 that takes into account the degree of erythema, induration/papulation, excoriation, and lichenification (each scored from 0 to 3 separately, half points are permitted) for each of four body regions, with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The severity of each sign is assessed using a 4-point scale (half points are permitted):
  * 0 = none
  * 1 = mild
  * 2 = moderate
  * 3 = severe A decrease in EASI indicates a positive outcome for the participant.
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle Cream | 1% DS107 Cream | 5% DS107 Cream
Number analyzed (Participants) | 106 | 110 | 110
score on a scale
  Week 2 | -3.14 (4.387) | -3.13 (5.390) | -2.72 (4.776)
  Week 4 | -6.19 (6.705) | -5.43 (6.358) | -5.57 (6.765)
  Week 6 | -7.28 (7.518) | -6.45 (7.198) | -7.40 (7.248)
  Week 10 | -8.47 (8.474) | -7.69 (7.143) | -8.74 (7.769)

6. Secondary Outcome: Proportion of Patients Achieving an Investigator's Global Assessment (IGA) Score of 0 (Clear) or 1 (Almost Clear) and a Decrease of at Least 2 Points in IGA in Treated Population Compared to Vehicle Population From Baseline to Week 2, 4, 6, 8, 10.
Description: Proportion of patients achieving an IGA score of 0 (clear) or 1 (almost clear) and a decrease of at least 2 points in IGA in treated population compared to vehicle population from baseline to Week 2, 4, 6, 8, 10. EASI quantifies the severity of a patient's atopic dermatitis (AD) based on both lesion severity and the percent of body surface area (BSA) affected. The EASI is a composite score ranging from 0-72 that takes into account the degree of erythema, induration/papulation, excoriation, and lichenification (each scored from 0 to 3 separately, half points are permitted) for each of four body regions, with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The severity of each sign is assessed using a 4-point scale (half points are permitted):
  * 0 = none
  * 1 = mild
  * 2 = moderate
  * 3 = severe A decrease in EASI indicates a positive outcome for the participant.
Time Frame: 10 weeks
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Vehicle Cream | 1% DS107 Cream | 5% DS107 Cream
Number analyzed (Participants) | 106 | 110 | 110
Proportion of participants
  Week 2 | 0.03 | 0.05 | 0.03
  Week 4 | 0.07 | 0.10 | 0.08
  Week 6 | 0.11 | 0.12 | 0.14
  Week 8 | 0.14 | 0.17 | 0.23
  Week 10 | 0.12 | 0.15 | 0.25

7. Secondary Outcome: Proportion of Patients Achieving a Decrease of at Least 2 Points in IGA in the Treated Populations Compared to Vehicle Population From Baseline to Week 2, 4, 6, 8, 10.
Description: Proportion of Patients Achieving a Decrease of at Least 2 Points in Investigator Global Assessment (IGA) in the Treated Populations Compared to Vehicle Population From Baseline to Week 2, 4, 6, 8, 10.
  The IGA scale awards a score of 0˗4 based on a 5-point severity scale from clear to severe disease (0 = clear, 1 = almost clear, 2 = mild disease, 3 = moderate disease, 4 = severe disease). IGA uses clinical characteristics of erythema, infiltration, papulation, and oozing/crusting as scoring guidelines for the overall severity assessment.
Time Frame: 10 weeks
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Vehicle Cream | 1% DS107 Cream | 5% DS107 Cream
Number analyzed (Participants) | 106 | 110 | 110
Proportion of participants
  Week 2 | 0.03 | 0.05 | 0.03
  Week 4 | 0.07 | 0.10 | 0.08
  Week 6 | 0.11 | 0.12 | 0.14
  Week 8 | 0.14 | 0.17 | 0.23
  Week 10 | 0.12 | 0.15 | 0.25

8. Secondary Outcome: Change From Baseline in IGA Score in the Treated Populations Compared to Vehicle Population at Weeks 2, 4, 6, 8, 10.
Description: The Global Investigator Assessment scale (IGA) scale awards a score of 0-4 based on a 5-point severity scale from clear to severe disease (0 = clear, 1 = almost clear, 2 = mild disease, 3
  = moderate disease, 4 = severe disease). The scale uses clinical characteristics of erythema, infiltration, papulation and oozing/crusting as scoring guidelines for the overall severity assessment. A decrease in IGA indicates a positive outcome for the participant.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8 and Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle Cream | 1% DS107 Cream | 5% DS107 Cream
Number analyzed (Participants) | 106 | 110 | 110
score on a scale
  Week 2 | -0.18 (0.562) | -0.27 (0.604) | -0.26 (0.585)
  Week 4 | -0.33 (0.719) | -0.57 (0.737) | -0.44 (0.709)
  Week 6 | -0.49 (0.840) | -0.70 (0.822) | -0.70 (0.827)
  Week 8 | -0.78 (0.871) | -0.85 (0.896) | -0.92 (0.953)
  Week 10 | -0.73 (0.881) | -0.80 (0.858) | -0.98 (0.987)

ADVERSE EVENTS:
Time Frame: Up to 10 weeks
Description: Any undesirable experience occurring to a patient who has signed the Informed Consent Form (ICF) and has taken their first dose of the study drug, whether or not considered related to the investigational Investigational Medicinal Product(s) (IMP). All Adverse Events (AEs) must be recorded in the case report form, defining relationship to IMP and severity.
Arm/Group | Vehicle Cream | 1% DS107 Cream | 5% DS107 Cream
All-Cause Mortality (participants affected / at risk) | 0/106 | 0/110 | 0/111
Serious Adverse Events (participants affected / at risk) | 1/106 | 1/110 | 0/111
Other Adverse Events (participants affected / at risk) | 38/106 | 48/110 | 40/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle Cream (N=106) | 1% DS107 Cream (N=110) | 5% DS107 Cream (N=111)
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle Cream (N=106) | 1% DS107 Cream (N=110) | 5% DS107 Cream (N=111)
Monocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 1 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus Hernia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Application Site Erythema (General disorders) | 0 | 1 | 1
Application Site Inflammation (General disorders) | 0 | 1 | 0
Application Site Pain (General disorders) | 1 | 2 | 4
Application Site Pruritus (General disorders) | 0 | 1 | 2
Application Site Reaction (General disorders) | 1 | 0 | 1
Application Site Swelling (General disorders) | 0 | 1 | 0
Influenza Like Illness (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 1
Peripheral Swelling (General disorders) | 1 | 0 | 0
Swelling (General disorders) | 0 | 1 | 0
Xerosis (General disorders) | 0 | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Dermatitis Infected (Infections and infestations) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0
Fungal Infection (Infections and infestations) | 0 | 1 | 0
Furuncle (Infections and infestations) | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 1
Helicobacter Zoster (Infections and infestations) | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 1
Impetigo (Infections and infestations) | 1 | 1 | 1
Infection (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 1 | 1
Otitis Media Acute (Infections and infestations) | 0 | 1 | 0
Perineal Infection (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Skin Bacterial Infection (Infections and infestations) | 1 | 0 | 0
Soft Tissue Infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 1
Tooth Abscess (Infections and infestations) | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 4 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 2 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 5 | 6 | 1
Arthropod Bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cataract Operation Complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Heat Stroke (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 1 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tooth Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood Creatine Phosphokinase (Investigations) | 0 | 1 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 1
Hepatic Enzyme Increased (Investigations) | 0 | 1 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Adenoma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Headache (Nervous system disorders) | 5 | 4 | 2
Migraine (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 2 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Tension Headache (Nervous system disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 4 | 5 | 2
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 4 | 5 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin Fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin Tightness (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Tonsillectomy (Surgical and medical procedures) | 1 | 0 | 0
Tooth Extraction (Surgical and medical procedures) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 2 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT02925793/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT02925793/SAP_001.pdf